CLINICAL TRIAL: NCT02918994
Title: LearningRx Cognitive Training for Traumatic Brain Injury (TBI): A Multiple Baseline Study Across Cases
Brief Title: LearningRx Cognitive Training for TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gibson Institute of Cognitive Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GICR-0916-B
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LearningRx cognitive training (Experimental): The intervention is a 60-hour, clinician-delivered cognitive training program.
  Interventions: Behavioral: LearningRx cognitive training

INTERVENTIONS:
Behavioral: LearningRx cognitive training — A clinician will deliver three 90-minute cognitive training sessions per week for 14 weeks. There are 16 different categories of leveled training procedures sequenced in intensity and difficulty for a total of 530 training tasks.

SUMMARY:
The purpose of this investigation is to conduct a series of case studies on the impact of LearningRx cognitive training on cognitive skills, brain structure, and daily functioning for participants with Traumatic Brain Injury (TBI).

DETAILED DESCRIPTION:
Using a multiple baseline design across cases with start point randomization, the proposed study will examine the outcomes from LearningRx one-on-one cognitive training across domains on standardized measures used to monitor treatment effectiveness for TBI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ previously diagnosed with TBI
* Living in the greater Colorado Springs area

Exclusion Criteria:

* No braces, metal implants, or claustrophobia that would contraindicate magnetic resonance imaging

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2018-10 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of overall cognitive function improvement | within 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Woodcock Johnson IV - Tests of Cognitive Abilities

SECONDARY OUTCOMES:
Evidence of change in brain activity | within 30 days after completing the intervention
  As confirmed by pretest to post-test changes in electrical activity measured by qEEG
Evidence of reduction in TBI symptoms | within 14 days after completing the intervention
  As confirmed by pretest to post-test changes on the Traumatic Brain Injury Checklist
Evidence of change in brain structure | within 30 days after completing the intervention
  Confirmed by change in pretest to post-test neuroimaging using MRI
Evidence of improvement in visual attention | with 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Conners Continous Performance Test (CPT-3)
Evidence of improvement in auditory attention | with 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Auditory Attention Test (CATA)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ledbetter, PhD, Principal Investigator — Gibson Institute of Cognitive Research; Amy L Moore, PhD, Study Director — Gibson Institute of Cognitive Research
Locations (1):
- Gibson Institute of Cognitive Research, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Will add to Harvard Dataverse

REFERENCES:
- [Derived] Moore AL, Carpenter DM 2nd, James RL, Miller TM, Moore JJ, Disbrow EA, Ledbetter CR. Neuroimaging and Neuropsychological Outcomes Following Clinician-Delivered Cognitive Training for Six Patients With Mild Brain Injury: A Multiple Case Study. Front Hum Neurosci. 2020 Jun 24;14:229. doi: 10.3389/fnhum.2020.00229. eCollection 2020. PMID 32670040